CLINICAL TRIAL: NCT01776268
Title: Effect of Colostrum on Innate Mucosal Immunity in Very Premature Infants
Brief Title: Effect of Colostrum on Mucosal Immunity in Very Low Birth Weight (VLBWs) Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, James Wynn, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 121760
Record Dates: First submitted 2013-01-17; First posted 2013-01-28 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Prematurity
Keywords: antimicrobial proteins
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral priming (Experimental): Mother's own colostrum is administered (0.1 mL to each cheek every 6 hours for 5 days) as soon as it is available from the mother regardless of when enteral feedings are initiated.
  Interventions: Other: Oral priming
- No oral priming (No Intervention): No oral priming

INTERVENTIONS:
Other: Oral priming — Mother's own colostrum is administered (0.1 mL to each cheek every 6 hours for 5 days) as soon as it is available from the mother regardless of when enteral feedings are initiated.
  Arms: Oral priming

SUMMARY:
Background:

Infection in preterm infants is a common, costly, and devastating problem frequently causing death or sequelae for survivors. An immature immune system underlies the frequency and severity of infections in this vulnerable population. The mouth is the site where microbes first meet the mucosal immune system. Antimicrobial proteins and peptides (APPs) in saliva kill microbes and improve immune cell function. Low APP levels increase the risk of developing infection. Colostrum and human milk reduce the risk of infection. This protective effect of human milk may come from supplying or stimulating infant production of APPs. No prior investigation has determined the concentration of APPs in saliva or the effect of human milk/formula on the APP concentrations in saliva.

Objective(s) and Hypothesis(es):

The investigators objectives are to identify and serially determine the concentrations of key APPs in colostrum, human milk, and preterm infant saliva using highly-sensitive and specific mass spectroscopy methods. The investigators study is designed to test the hypotheses that (a) all saliva APPs increase over time, (b) APP concentrations are higher in colostrum as compared to human milk, and (c) APPs are increased in saliva of infants that receive colostrum orally compared to those that do not.

Potential Impact:

If increased saliva APP levels are associated with oral colostrum priming, this discovery would advance understanding of the immune properties of human milk and identify oral APPs as important immune elements and potential therapeutic targets in this vulnerable population. This knowledge has the potential to alter feeding practices and provide a safe, low cost means to improve immune function and significantly improve outcomes for preterm infants.

DETAILED DESCRIPTION:
Background: Between 20 and 60% of very low birth weight (VLBW) infants are diagnosed with infection during their initial hospitalization2-9. Infection in preterm infants is a costly and devastating problem associated with high mortality and debilitating survivor morbidity. High infection rates are attributed to suboptimal preterm neonatal immune function. In depth investigation of the unique properties of the preterm neonatal immune function is necessary to identify novel interventions that can translate into improved neonatal outcomes.

Mucosal surfaces are critical immune barriers that shield against host microbial invasion by surface-colonizing commensal or potentially pathogenic organisms. Antimicrobial proteins and peptides (APPs) on mucosal surfaces reduce microbial burden individually and synergistically by direct killing of microbes and by improving immune surveillance through activation of local sentinel cells. Deficiencies in these innate immune proteins predispose the host to infection or dysregulated inflammation. Two major classes of APPs (defensins and cathelicidin) are present on mucosal surfaces in adults. Colostrum and human milk (HM) contain some APPs that may play an adjuvant role on mucosal sites including the mouth. HM ingestion is associated with a decreased risk of developing sepsis and necrotizing enterocolitis in preterm infants. One potential mechanism behind the reduction in infection risk associated with HM feeding may be enhanced immunocompetence through provision of APPs and induction of neonatal APP production. Investigators are not aware of any investigation that has determined the neonatal salivary concentration of any APP or the effect of oral priming (OP) with colostrum on the concentration of salivary APPs. It is also unknown whether OP with formula modifies salivary APPs.

Objectives and Hypotheses: Our objectives are to determine: 1) the concentration of salivary APPs from preterm infants at baseline and 7 days later, 2) the effect of oral priming (OP) with either human milk or formula on salivary APP concentrations, and 3) the concentration of APPs in colostrum as compared to milk. Our hypotheses are: 1) All salivary APPs increase over time in preterm infants (with or without OP) 2) Compared with formula OP or no OP, colostrum OP is associated with a significantly greater increase in salivary LL-37 and hBD2 concentrations and 3) Colostrum contains a greater concentration of LL-37 compared to human milk.

Design: Following the mother's decision to provide human milk or formula to her preterm newborn, VLBW infants will be randomized to receive OP or not. Investigators will compare the concentration of salivary APPs from VLBW infants that receive OP to VLBW infants that do not. Saliva will be sampled prior to and after 5 days of OP. Time-matched saliva samples will be obtained from the infants that do not receive OP. APP concentrations will be compared between the biological mother's colostrum (both whey and fat fractions) and her transitional milk (produced >7 days after birth). To account for the heterogeneous VLBW population, investigators will study 200 infants (50 infants/group, 4 groups) to test our hypotheses. Both inborn and outborn VLBW infants are eligible. Exclusion criteria include infants with a medical contraindication for oral or enteral feeds, congenital anomalies or chromosomal disorders. Saliva and milk-based proteomes including APPs will be determined using Matrix Assisted Laser Desorption/Ionization Time-of-Flight (MALDI-TOF).

Potential Impact: This is the first study of APPs in saliva of human neonates. If increased saliva APP levels are associated with colostrum OP, this discovery would add to our understanding of the immune properties of human milk. Identification of APPs as important elements that improve immune function is likely to alter the approach to infant nutrition and improve outcomes for premature infants. Ultimately, our goal is to determine whether there is an association between APP levels in neonatal saliva and the incidence of neonatal infection (including NEC) in an appropriately powered clinical study based on the data generated in this proposal.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight (<1500 g)
* Gestational age <30 weeks
* Admission to NICU (born at Vanderbilt or transferred in for care)
* English or Spanish-speaking parents

Exclusion Criteria:

* Does not meet inclusion criteria
* Parent does not give study consent
* Has congenital anomalies, chromosomal disorder or medical contraindication to oral/enteral feedings

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Wynn, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Monroe Carell Jr Children's Hospital at Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Romano-Keeler J, Azcarate-Peril MA, Weitkamp JH, Slaughter JC, McDonald WH, Meng S, Latuga MS, Wynn JL. Oral colostrum priming shortens hospitalization without changing the immunomicrobial milieu. J Perinatol. 2017 Jan;37(1):36-41. doi: 10.1038/jp.2016.161. Epub 2016 Sep 29. PMID 27684425
- See also: Oral colostrum priming shortens hospitalization without changing the immunomicrobial milieu — http://www.nature.com/jp/journal/v37/n1/full/jp2016161a.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Colostrum Priming: Intervention:Mother's own colostrum is administered (0.1 mL to each cheek every 6 hours for 5 days) as soon as it is available from the mother regardless of when enteral feedings are initiated.
Period: Overall Study
Arm/Group | Colostrum Priming | no Oral Priming
Started | 48 | 51
Completed | 48 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oral Priming: Intervention:Mother's own colostrum is administered (0.1 mL to each cheek every 6 hours for 5 days) as soon as it is available from the mother regardless of when enteral feedings are initiated.
- no Oral Priming: No oral priming: no intervention
- Total: Total of all reporting groups
Arm/Group | Oral Priming | no Oral Priming | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Continuous [Mean (Inter-Quartile Range); unit: weeks] — Gestational age in weeks
  weeks | 30 [27 to 31] | 29 [28 to 30] | 29 [27 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 30 | 54
  Male | 24 | 21 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Mother's Ethnicity is reported
  Participants
    Hispanic or Latino | 8 | 7 | 15
    Not Hispanic or Latino | 40 | 44 | 84
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Mother's Race is reported
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 19 | 13 | 32
    White | 28 | 35 | 63
    More than one race | 1 | 2 | 3
    Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 48 | 51 | 99
Birth Weight [Mean (Inter-Quartile Range); unit: grams] | 1272 [988 to 1602] | 1170 [905 to 1340] | 1219 [905 to 1602]
APGAR [Mean (Inter-Quartile Range); unit: units on a scale] — APGAR 0=worst 10=best Activity, Pulse, Grimace, Appearance, and Respiration.
  Activity 0 Limp
  1. Some flexion of arms and legs
  2. Active motion
  Pulse 0 No heart rate
  1. <100 beats per minute
  2. At least 100 beats/minute
  Grimace during suctioning 0 No response
  1. Grimace
  2. Grimace and pull away, cough
  Appearance 0 whole body bluish-gray or pale
  1. Good color in body with bluish hands or feet
  2. Good color all over
  Respiration 0 Not breathing
  1. Weak cry; , slow or irregular breathing
  2. Good, strong cry; normal rate and effort of breathing
  units on a scale | 7 [6 to 8] | 7 [6 to 8] | 7 [6 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Concentration of APPs Before Oral Priming
Description: Saliva will be sampled on day 1-2 of life prior to oral priming. Investigators are assessing saliva for a change in the concentration of antimicrobial proteins.
Time Frame: days 1-2 of life
Measure: Mean (Inter-Quartile Range); unit: femtomole (fmol)
Arm/Group | Oral Priming | No Oral Priming
Number analyzed (Participants) | 48 | 51
femtomole (fmol)
  S100a7-S1 | 17 [8 to 39] | 22 [7 to 45]
  S100a7-S2 | 35 [5 to 60] | 42 [5 to 169]
  S100a8-S1 | 101 [39 to 313] | 102 [49 to 305]
  S100a8-S2 | 495 [190 to 854] | 683 [109 to 1064]
  S100a9-S1 | 1669 [755 to 2540] | 2392 [287 to 3465]
  S100a9-S2 | 198 [112 to 337] | 364 [67 to 614]
  Surfactant protein A | 5 [0 to 5] | 0 [0 to 7]
  α-Defensin 1-S1 | 1 [0 to 1] | 1 [0 to 3]
  α-Defensin 5 | 1 [1 to 1] | 1 [1 to 7]
  Lactoferrin-S1 | 11 [1 to 23] | 15 [1 to 40]
  Lactoferrin-S2 | 10 [7 to 17] | 14 [8 to 20]
  Immunoglobulin A | 10 [10 to 196] | 10 [10 to 68]
  Lysozyme C-S1 | 1257 [698 to 2184] | 1122 [559 to 2058]
  Lysozyme C-S2 | 0 [0 to 12] | 0 [0 to 20]

2. Primary Outcome: Concentration of APPs After Oral Priming
Description: Saliva will be sampled 24-48 hours after the 5-days of oral priming is completed. Investigators are assessing saliva for a change in the concentration of antimicrobial proteins.
Time Frame: days 7-9 of life
Measure: Mean (Inter-Quartile Range); unit: femtomole (fmol)
Arm/Group | Oral Priming | No Oral Priming
Number analyzed (Participants) | 48 | 51
femtomole (fmol)
  S100a7-S1 | 15 [8 to 27] | 20 [9 to 28]
  S100a7-S2 | 18 [5 to 68] | 38 [5 to 88]
  S100a8-S1 | 144 [44 to 308] | 206 [57 to 457]
  S100a8-S2 | 511 [197 to 789] | 562 [252 to 1037]
  S100a9-S1 | 1777 [934 to 2473] | 1886 [731 to 4008]
  S100a9-S2 | 241 [114 to 311] | 319 [114 to 498]
  Surfactant protein A | 0 [0 to 5] | 5 [0 to 6]
  α-Defensin 1-S1 | 1 [0 to 5] | 1 [0 to 10]
  α-Defensin 5 | 1 [0 to 1] | 1 [0 to 1]
  Lactoferrin-S1 | 57 [1 to 92] | 29 [1 to 91]
  Lactoferrin-S2 | 49 [14 to 103] | 21 [12 to 38]
  Immunoglobulin A | 102 [29 to 1373] | 42 [10 to 328]
  Lysozyme C-S1 | 1680 [836 to 3416] | 1972 [1344 to 2617]
  Lysozyme C-S2 | 15 [0 to 31] | 8 [0 to 23]

ADVERSE EVENTS:
Arm/Group | Oral Priming | no Oral Priming
All-Cause Mortality (participants affected / at risk) | 1/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/48 | 0/51
Other Adverse Events (participants affected / at risk) | 0/48 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Priming (N=48) | no Oral Priming (N=51)
Death (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes